CLINICAL TRIAL: NCT00569803
Title: Pharmacokinetics, Safety and Immunogenicity of Single Doses of Belatacept Administered Subcutaneously to Healthy Subjects
Brief Title: Subcutaneous Pharmacokinetics of Belatacept
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IM103-046
Record Dates: First submitted 2007-11-30; First posted 2007-12-07 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Transplantation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Belatacept 50 mg Subcutaneous Injection (Active Comparator): Belatacept 50 mg subcutaneous (SC) injection
  Interventions: Drug: belatacept
- Belatacept 100 mg Subcutaneous Injection (Active Comparator): Belatacept 100 mg SC injection
  Interventions: Drug: belatacept
- Belatacept 125 mg Subcutaneous Injection (Active Comparator): Belatacept 125 mg SC injection
  Interventions: Drug: belatacept
- Belatacept 150 mg Subcutaneous Injections (Active Comparator): 2 SC injections of 75 mg Belatacept
  Interventions: Drug: belatacept
- Belatacept 200 mg Subcutaneous Injections (Active Comparator): 2 SC injections of 100 mg Belatacept
  Interventions: Drug: belatacept
- Belatacept 250 mg Subcutaneous Injections (Active Comparator): 2 SC injections of 125 mg Belatacept
  Interventions: Drug: belatacept
- Belatacept 125 mg Intravenous Infusion (Active Comparator): 125 mg Belatacept intravenous (IV) injection
  Interventions: Drug: belatacept
- Placebo (Placebo Comparator): SC injection of placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: belatacept — single dose, 116 days
  Arms: Belatacept 100 mg Subcutaneous Injection; Belatacept 125 mg Intravenous Infusion; Belatacept 125 mg Subcutaneous Injection; Belatacept 150 mg Subcutaneous Injections; Belatacept 200 mg Subcutaneous Injections; Belatacept 250 mg Subcutaneous Injections; Belatacept 50 mg Subcutaneous Injection
Drug: Placebo — Subcutaneous injection of placebo solution (product ID: 224818-N000- 029)
  Arms: Placebo

SUMMARY:
Pharmacokinetics, Bioavailability, Safety and Immunogenicity of Single Doses of Belatacept Administered Subcutaneously to Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 65 years old
* Subjects must weigh less than or equal to 100 kg

Exclusion Criteria:

* Inability to tolerate injections or IV infusions
* autoimmune disorders
* TB
* herpes
* HCV
* HBV
* HIV
* bacterial or viral infection
* history of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 153 participants were enrolled, with 106 discontinuing prior to study drug administration because they no longer met study criteria or they withdrew consent. 47 participants met all eligibility criteria and received study medication. 1 subject, who received an incomplete dose due to an injection syringe leak, was replaced.
Groups:
- Belatacept 50 mg Subcutaneous Injection: Belatacept 50 mg subcutaneous (SC) injection into anterior thigh, 0.4 mL injection volume
- Belatacept 100 mg Subcutaneous Injection: Belatacept 100 mg SC injection into anterior thigh, 0.8 mL injection volume
- Belatacept 125 mg Subcutaneous Injection: Belatacept 125 mg SC injection into anterior thigh, 1.0 mL injection volume
- Belatacept 150 mg Subcutaneous Injections: Participants received 2 SC injections of 75 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
- Belatacept 200 mg Subcutaneous Injections: Participants received 2 SC injections of 100 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
- Belatacept 250 mg Subcutaneous Injections: Participants received 2 SC injections of 125 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
Period: Overall Study
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Started | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
Completed | 4 | 5 | 5 | 5 | 5 | 5 | 10 | 5
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — injection syringe leaked during dosing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (11) | 27 (12) | 28 (12) | 34 (18) | 31 (11) | 31 (10) | 32 (16) | 27 (6) | 30 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 2 | 3 | 2 | 2 | 4 | 21
  Male | 1 | 3 | 3 | 4 | 2 | 3 | 8 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Belatacept
Description: Maximum observed serum concentration (Cmax) values were derived from serum concentration versus time data and reported in micrograms per milliliter (ug/mL).
Time Frame: Immediately before dose, 0.5, 2, 6, 12, 24, 36, 48, 60, 72, 84 hours post-dose, Days 5, 6, 7, 8, 14, 21, 28, 35, 42, 56, 86 and 116
Population: All participants treated with Belatacept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 10
ug/mL | 3.9 (30) | 6.2 (34) | 8.5 (50) | 11.1 (19) | 14.5 (16) | 14.5 (18) | 42.4 (16)

2. Primary Outcome: Time of Maximum Observed Serum Concentration (Tmax) of Belatacept
Description: Time of maximum observed serum concentration (Tmax) values were derived from serum concentration versus time data for all participants treated with Belatacept.
Time Frame: as for outcome 1
Population: All participants treated with Belatacept
Measure: Median (Full Range); unit: hours
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 10
hours | 84 [36 to 96] | 60 [48 to 120] | 96 [48 to 144] | 60 [36 to 96] | 60 [24 to 84] | 72 [60 to 96] | 0.5 [0.2 to 2.0]

3. Primary Outcome: Adjusted Geometric Means of Area Under the Serum Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC(0-T)) for Belatacept
Description: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T)) was derived from serum concentration versus time data. Adjusted geometric means were reported in microgram hours per milliliter (ug*h/mL).
Time Frame: as for outcome 1
Population: All participants treated with Belatacept
Measure: Geometric Mean (90% Confidence Interval); unit: ug*h/mL
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 10
ug*h/mL | 2587 [2132 to 3139] | 1848 [1523 to 2242] | 2371 [1954 to 2876] | 2703 [2228 to 3280] | 2650 [2184 to 3215] | 2193 [1807 to 2660] | 3023 [2637 to 3466]
Statistical Analysis 1: Comparison: Belatacept 50 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.86, 90% CI 2-sided [0.68 to 1.08] — Ratio of Geometric Means: 50mg SC over 125mg IV
Statistical Analysis 2: Comparison: Belatacept 100 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.61, 90% CI 2-sided [0.48 to 0.77] — Ratio of Geometric Means: 100mg SC over 125mg IV
Statistical Analysis 3: Comparison: Belatacept 125 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.78, 90% CI 2-sided [0.62 to 0.99] — Ratio of Geometric Means: 125mg SC over 125mg IV
Statistical Analysis 4: Comparison: Belatacept 150 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.89, 90% CI 2-sided [0.71 to 1.13] — Ratio of Geometric Means: 150mg SC over 125mg IV
Statistical Analysis 5: Comparison: Belatacept 200 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.88, 90% CI 2-sided [0.69 to 1.11] — Ratio of Geometric Means: 200mg SC over 125mg IV
Statistical Analysis 6: Comparison: Belatacept 250 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.73, 90% CI 2-sided [0.57 to 0.92] — Ratio of Geometric Means: 250mg SC over 125mg IV

4. Primary Outcome: Adjusted Geometric Means of Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) for Belatacept
Description: Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) was derived from serum concentration versus time data. Adjusted geometric means were reported in microgram hours per milliliter (ug*h/mL)
Time Frame: as for outcome 1
Population: All participants treated with Belatacept
Measure: Geometric Mean (90% Confidence Interval); unit: ug*h/mL
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 10
ug*h/mL | 2639 [2172 to 3205] | 1851 [1524 to 2248] | 2380 [1959 to 2891] | 2719 [2238 to 3303] | 2666 [2194 to 3238] | 2201 [1812 to 2673] | 3031 [2642 to 3478]
Statistical Analysis 1: Comparison: Belatacept 50 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.87, 90% CI 2-sided [0.69 to 1.10] — Ratio of Geometric Means: 50mg SC over 125mg IV
Statistical Analysis 2: Comparison: Belatacept 100 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.61, 90% CI 2-sided [0.48 to 0.77] — Ratio of Geometric Means: 100mg SC over 125mg IV
Statistical Analysis 3: Comparison: Belatacept 125 mg Subcutaneous Injection vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.79, 90% CI 2-sided [0.62 to 1.00] — Ratio of Geometric Means: 125mg SC over 125mg IV
Statistical Analysis 4: Comparison: Belatacept 150 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.90, 90% CI 2-sided [0.71 to 1.14] — Ratio of Geometric Means: 150mg SC over 125mg IV
Statistical Analysis 5: Comparison: Belatacept 200 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.88, 90% CI 2-sided [0.69 to 1.12] — Ratio of Geometric Means: 200mg SC over 125mg IV
Statistical Analysis 6: Comparison: Belatacept 250 mg Subcutaneous Injections vs Belatacept 125 mg Intravenous Infusion; Test type: Superiority or Other; Ratio of Geometric Means = 0.73, 90% CI 2-sided [0.57 to 0.92] — Ratio of Geometric Means: 250mg SC over 125mg IV

5. Primary Outcome: Serum Half-life (T-HALF) of Belatacept
Description: Serum half-life (T-HALF) was determined from serum concentration versus time data and was reported in hours.
Time Frame: as for outcome 1
Population: All participants treated with Belatacept
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 10
hours | 112 (25.7) | 100 (10.1) | 135 (47.6) | 158 (46.9) | 161 (45.3) | 150 (43.6) | 130 (27.6)

6. Primary Outcome: Apparent Total Body Clearance (CLT/F) of SC Belatacept
Description: Apparent total body clearance (CLT/F) was derived from serum concentration versus time data for all participants who received subcutaneous (SC) Belatacept injections. Units reported in milliliters per hour (mL/h).
Time Frame: as for outcome 1
Population: All participants treated with SC Belatacept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
mL/h | 47.4 (27) | 67.5 (34) | 52.5 (31) | 46.0 (26) | 46.9 (21) | 56.8 (20)

7. Primary Outcome: Total Body Clearance (CLT) of IV Belatacept
Description: Total body clearance (CLT) was derived from serum concentration versus time data for all participants that were treated with IV Belatacept. Units reported in milliliters per hour (mL/h)
Time Frame: as for outcome 1
Population: All participants treated with IV Belatacept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 10
mL/h | 41.2 (21)

8. Primary Outcome: Volume of Distribution at Steady State (VSS) for IV Belatacept
Description: Volume of distribution at steady state (VSS) was derived from serum concentration versus time data for all participants treated with IV Belatacept.
Time Frame: as for outcome 1
Population: All participants treated with IV Belatacept
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 10
Liters | 7.3 (1.27)

9. Primary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) for SC Belatacept
Description: Apparent volume of distribution at steady state (Vss/F) was derived from concentration versus time data for all participants treated with subcutaneous (SC) Belatacept.
Time Frame: as for outcome 1
Population: All participants treated with SC Belatacept
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Liters | 10.79 (31.02) | 15.30 (28.79) | 14.12 (36.63) | 12.75 (14.20) | 13.34 (13.77) | 15.82 (11.92)

10. Secondary Outcome: Effect of Number of Injection Sites on Subcutaneous Belatacept Absorption
Description: AUC(0-T) and AUC(INF) for Belatacept were derived from serum concentration versus time data to assess the effect of number of injection sites on the subcutaneous absorption of Belatacept. All treatments were dose-normalized to 50mg. Adjusted geometric means reported in microgram hours per milliliter (ug*h/mL).
  AUC(0-T) = Area Under the Serum Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration.
  AUC(INF) = Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinite Time.
Time Frame: as for outcome 1
Population: All participants treated with Belatacept
Measure: Geometric Mean (90% Confidence Interval); unit: ug*h/mL
Groups:
- 1 Injection Site: Participants receiving treatments of 50mg, 100mg and 125mg Subcutaneous Belatacept were injected at 1 site at the anterior thigh.
- 2 Injection Sites: Participants receiving treatments of 150mg, 200mg and 250mg Subcutaneous Belatacept were injected at 2 sites; one injection equal to half the total dose was delivered to the anterior thigh on each side.
Arm/Group | 1 Injection Site | 2 Injection Sites
Number analyzed (Participants) | 15 | 15
ug*h/mL
  AUC(0-T) | 898 [794 to 1017] | 1002 [885 to 1134]
  AUC(INF) | 906 [799 to 1027] | 1007 [888 to 1142]
Statistical Analysis 1: Comparison: 1 Injection Site vs 2 Injection Sites; Test type: Superiority or Other; Ratio of Geometric Means = 0.90, 90% CI 2-sided [0.75 to 1.07] — AUC(0-T) Ratio of Geometric Means: 1 injection site over 2 injection sites
Statistical Analysis 2: Comparison: 1 Injection Site vs 2 Injection Sites; Test type: Superiority or Other; Ratio of Geometric Means = 0.90, 90% CI 2-sided [0.75 to 1.07] — AUC(INF) Ratio of Geometric Means: 1 injection site over 2 injection sites

11. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital signs (body temperature, respiratory rate, seated blood pressure, and heart rate) were recorded at screening. All significant findings were evaluated by the investigator, and all abnormalities were listed.
Time Frame: 1 day pre-dose, Days 1, 2, 5, 14, 28, 42, 86 and 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Participants were assessed for erythema, heat, pain, pruritis and swelling at the injection sites and were characterized by the investigator as mild, moderate or severe reactions.
Time Frame: 0.5, 2, 6 and 24 hours post-dose, Days 3, 4, 5, 6, 7, 8, 14, 21 and 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants
  mild reaction | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  moderate reaction | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  severe reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: All clinically significant deviations from normal physical examinations were reported.
Time Frame: Days 1, 2, 5, 14, 28, 42, 86, 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Participants underwent a 12-lead ECG assessment at Screening (Day 1) and Study Discharge (Day 116). All investigator-assessed ECG abnormalities were reported.
Time Frame: Days 1 and 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants
  Screening (Day 1) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
  Study Discharge (Day 116) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0

15. Secondary Outcome: Number of Participants With Marked Hematology Laboratory Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities:
  Hemoglobin (grams per deciliter:g/dL): <0.85*Pre-Rx. Hematocrit (%): <0.85*Pre-Rx. Platelet Count (*10^9 cells per liter:c/L): <0.85*LLN or >1.5*ULN (if Pre-Rx<LLN, use <0.85*Pre-Rx).
  Leukocytes (*10^3 cells per microliter: c/uL): <0.9*LLN, >1.2*ULN (if Pre-Rx<LLN, use <0.85*Pre-Rx or >ULN, if Pre-Rx>ULN, use >1.15*Pre-Rx or <LLN) Neutrophils+Bands (*10^3 c/uL): <=1.500. Lymphocytes (*10^3 c/uL): <0.750 or >7.500. Monocytes (*10^3 c/uL): >2.000. Basophils (*10^3 c/uL): >0.400. Eosinophils (*10^3 c/uL): >0.750.
Time Frame: Day 1 Pre-dose, Days 2, 5, 14, 28, 42, 86, 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants
  Hemoglobin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils + Bands (absolute) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Lymphocytes (absolute) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Monocytes (absolute) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (absolute) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (absolute) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Marked Serum Chemistry Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities:
  Alkaline Phosphatase (units per liter: U/L), Aspartate Aminotransferase (U/L), Alanine Aminotransferase (U/L): >1.25*ULN (if Pre-Rx>ULN, use >1.25*Pre-Rx).
  Bilirubin (milligrams per deciliter: mg/dL): >1.1*ULN (if Pre-Rx>ULN, use >1.25*Pre-Rx).
  Blood Urea Nitrogen (mg/dL): >1.1*ULN (if Pre-Rx>ULN, use >1.2*Pre-Rx). Creatinine (mg/dL): >1.33*Pre-Rx. Sodium (milliequivalents per Liter: mEq/L): <0.95*LLN, >1.05*ULN (if Pre-Rx<LLN: <0.95*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.05*Pre-Rx, <LLN).
  Potassium(mEq/L), Chloride (mEq/L), Calcium(mg/dL): <0.9*LLN, >1.1*ULN (if Pre-Rx<LLN: <0.9*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.1*Pre-Rx, <LLN).
  Phosphorus (mg/dL): <0.85*LLN, >1.25*ULN (if Pre-Rx<LLN, <0.85*Pre-Rx, >ULN. if Pre-Rx>ULN: >1.25*Pre-Rx, <LLN).
Time Frame: Day 1 Pre-dose, Days 2, 5, 14, 28, 42, 86, 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants
  Alkaline Phosphatase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Alanine Aminotransferase | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Bilirubin | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Blood Urea Nitrogen | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, Serum | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, Serum | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Chloride, Serum | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, Total | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorus, Inorganic | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: LLN=Lower Limit of Normal, ULN=Upper Limit of Normal, Pre-Rx=Value before first dose. Lab values that met the following criteria were marked as abnormalities:
  Glucose (mg/dL): <0.8*LLN, >1.5*ULN (if Pre-Rx<LLN: <0.8*Pre-Rx, >ULN. If Pre-Rx>ULN: >2.0*Pre-Rx, <LLN).
  Protein (grams per deciliter: g/dL): <0.9*LLN, >1.1*ULN (if Pre-Rx<LLN: <0.9*Pre-Rx, >ULN. If Pre-Rx>ULN: >1.1*Pre-Rx, <LLN).
  Albumin (g/dL): <0.9*LLN (if Pre-Rx<LLN: <0.9*Pre-Rx). Uric Acid (mg.dL): >1.2*ULN (if Pre-Rx>ULN: >1.25*Pre-Rx). Lactate Dehydrogenase (U/L): >1.25*ULN (if Pre-Rx>ULN: >1.5*Pre-Rx)
Time Frame: Day 1 Pre-dose, Days 2, 5, 14, 28, 42, 86, 116
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10 | 6
participants
  Glucose, Fasting Serum | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Protein, Total | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Uric Acid | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Positive Immunogenicity to Belatacept
Description: The number of participants with positive immunogenicity to Belatacept was reported for each arm. Positive immunogenicity was defined as the presence of a positive antibody response generated against Belatacept.
Time Frame: Days 1, 14, 28, 42, 56, 86, 116
Population: All participants treated with Belatacept
Measure: Number; unit: participants
Arm/Group | Belatacept 50 mg Subcutaneous Injection | Belatacept 100 mg Subcutaneous Injection | Belatacept 125 mg Subcutaneous Injection | Belatacept 150 mg Subcutaneous Injections | Belatacept 200 mg Subcutaneous Injections | Belatacept 250 mg Subcutaneous Injections | Belatacept 125 mg Intravenous Infusion
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5 | 10
participants | 4 | 5 | 5 | 5 | 5 | 5 | 10

ADVERSE EVENTS:
Time Frame: From Day 1 until 30 days post discontinuation of dosing, up to August 2008 (approximately 8 months)
Description: Study initiated: December 2007
  Study completed: August 2008
  Participants underwent regularly scheduled investigator assessments and clinical laboratory evaluations as described in the study protocol.
Groups:
- Belatacept 50mg SC: Belatacept 50 mg subcutaneous (SC) injection into anterior thigh, 0.4 mL injection volume
- Belatacept 100mg SC: Belatacept 100 mg SC injection into anterior thigh, 0.8 mL injection volume
- Belatacept 125mg SC: Belatacept 125 mg SC injection into anterior thigh, 1.0 mL injection volume
- Belatacept 150mg SC: Participants received 2 SC injections of 75 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
- Belatacept 200mg SC: Participants received 2 SC injections of 100 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
- Belatacept 250mg SC: Participants received 2 SC injections of 125 mg Belatacept each, in the anterior thighs. One injection was given in each thigh, with the second injection immediately following the first injection.
- Belatacept 125mg IV: 125 mg Belatacept intravenous (IV) injection
- All Belatacept: All participants treated with IV or SC Belatacept of any dose
Arm/Group | Belatacept 50mg SC | Belatacept 100mg SC | Belatacept 125mg SC | Belatacept 150mg SC | Belatacept 200mg SC | Belatacept 250mg SC | Belatacept 125mg IV | PLACEBO | All Belatacept
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/5 | 0/10 | 0/6 | 0/41
Other Adverse Events (participants affected / at risk) | 2/5 | 3/5 | 3/5 | 4/6 | 2/5 | 2/5 | 7/10 | 1/6 | 23/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept 50mg SC (N=5) | Belatacept 100mg SC (N=5) | Belatacept 125mg SC (N=5) | Belatacept 150mg SC (N=6) | Belatacept 200mg SC (N=5) | Belatacept 250mg SC (N=5) | Belatacept 125mg IV (N=10) | PLACEBO (N=6) | All Belatacept (N=41)
Headache (Nervous system disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 3 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 8
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.